CLINICAL TRIAL: NCT04298086
Title: Pharmacodynamic Response to Exercise Treatment and Plant-Based Diet in Overweight/Obese Postmenopausal Women With Primary Hormone Receptor Positive Breast Cancer: A Phase 2 Randomized Control Trial
Brief Title: A Study of the Body's Response to Exercise and a Plant-Based Diet in Overweight Postmenopausal Women With Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other); McGill University (Other); University of Kansas Medical Center (Other); Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-486
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Primary Hormone Receptor Positive Breast Cancer
Keywords: Postmenopausal Women; Overweight/Obese; Plant-Based Diet; 19-486
MeSH Terms: conditions — Breast Neoplasms; Overweight; Obesity | interventions — Diet, Plant-Based; Exercise

STUDY DESIGN:
Intervention Model Description: A single-center, phase 2 randomized control trial of structured exercise treatment and plant-based diet versus physical activity and nutrition counseling for 24 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Treatment and Plant-Based Diet (Experimental): Will consist of structured exercise treatment plus a calorie-restricted plant-based diet. Exercise treatment will consist of individualized walking delivered up to 7 times weekly to achieve the patient-specific goal energy expenditure. Training sessions will be performed on a treadmill under remote surveillance using a telemedicine approach (i.e.,TeleEx) established in the Exercise-Oncology (ExOnc) Service. Pre-prepared meals, including 6 dinners and 6 lunches per week, will be shipped to the partipant's home during the intervention. If a patient is temporarily unable to complete supervised sessions as a result of unforeseen circumstances, patients may be assigned low intensity unsupervised training sessions per EP/PI discretion
  Interventions: Other: Exercise Treatment; Other: Plant-Based Diet; Other: Replication Exercise Test
- Physical activity and nutrition counseling (Active Comparator): Patients will receive a home-based, general physical activity program and nutrition counseling. Specifically, all patients assigned to the counseling arm will receive a study kit which includes an activity tracker, heart rate monitor, scale, and tablet. Treadmills may also be provided to patients in the counseling arm if they do not already have access to one.
  Interventions: Other: Physical activity; Other: Nutrition counseling

INTERVENTIONS:
Other: Exercise Treatment — Exercise treatment will consist of individualized walking delivered up to 7 times weekly to achieve the patient-specific goal energy expenditure. Training sessions will be performed on a treadmill at under remote surveillance using a telemedicine approach (i.e.,TeleEx) established in the Exercise-Oncology (ExOnc) Service.
  Arms: Exercise Treatment and Plant-Based Diet
Other: Plant-Based Diet — Pre-prepared meals, including 6 dinners and 6 lunches per week, will be shipped to the partipant's home during the intervention.
  Arms: Exercise Treatment and Plant-Based Diet
Other: Physical activity — Treadmills and low-calorie recipes will be provided to patients in the counseling arm.
  Arms: Physical activity and nutrition counseling
Other: Nutrition counseling — Nutrition program including regular counseling by exercise physiologists and registered dieticians (RDs).
  Arms: Physical activity and nutrition counseling
Other: Replication Exercise Test — Exercise capacity will be reassessed by a replication exercise test at week 6 in the intervention group only.
  Arms: Exercise Treatment and Plant-Based Diet

SUMMARY:
The purpose of this study is to find out what effects, if any, exercise and a plant-based diet have on aromatase levels in postmenopausal women who are overweight and being treated with an aromatase inhibitor for their HR+ breast cancer. The study will also look at other ways diet and exercise may affect your body (for example, changing the way your breast tissue expresses or makes genes) and your quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed, HR-positive (ER and/or PR) stage 1-3 breast cancer
* Completed anti-HER2 therapy, if HER2-positive
* Postmenopausal status defined by lack of menses for 2 years, oophorectomy, or medical ovarian suppression
* At least 3 months post completion of chemotherapy, if administered
* At least 3 months post radiation, if administered
* Receiving adjuvant endocrine therapy with an aromatase inhibitor (anastrozole, letrozole, exemestane)
* ECOG performance status of 0 to 1
* Sedentary (i.e.,performing <150 minutes / week of exercise structured moderate-intensity or strenuous-intensity)
* Age ≥ 18
* BMI ≥ 27
* Able to achieve an acceptable peak baseline CPET, as defined by any of the following criteria and in the absence of high risk ECG findings or other inappropriate response to exercise as determined by the investigator:

  * Achieved a plateau in oxygen consumption, concurrent with an increase in power output
  * A respiratory exchange ratio ≥ 1.10
  * Attainment of maximal predicted heart rate (HRmax) (i.e., within10 bpm of age- predicted HRmax [HRmax= 220 - Age (years)]
  * Volitional exhaustion, as measured by a rating of perceived exertion (RPE) ≥ 18 on the BORG scale.
* Willingness to comply with all study-related procedures
* Intact breast available for biopsy

Exclusion Criteria:

* Presence of metastatic disease
* Any concurrent malignancy requiring active treatment with the exception of selective estrogen receptor modulators and aromatase inhibitors
* Insulin-dependent diabetes mellitus or non-insulin dependent diabetes mellitus on insulin therapy
* Enrollment onto any other interventional investigational study except interventions determined by the PI not to confound the effect of exercise or diet on study outcomes
* Mental impairment leading to inability to cooperate
* Any of the following contraindications to exercise:

  1. Acute myocardial infarction within 3-5 days of any planned study procedures;
  2. Unstable angina
  3. Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
  4. Recurrent syncope
  5. Active endocarditis
  6. Acute myocarditis or pericarditis
  7. Symptomatic severe aortic stenosis
  8. Uncontrolled heart failure
  9. Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures
  10. Thrombosis of lower extremities
  11. Suspected dissecting aneurysm
  12. Uncontrolled asthma
  13. Pulmonary edema
  14. Respiratory failure
  15. Acute non-cardiopulmonary disorders that may affect exercise performance
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the subject a poor candidate for study participation.
* Nut or legume allergy
* Concurrent participation in weight loss programs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 43 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
change in breast aromatase levels | 24 weeks post-intervention
  Will explore the data using descriptive statistics and graphical methods, such as summarizing the aromatase levels at baseline and at 24 weeks using means and medians and plotting the data to visualize changes over time. To compare the aromatase levels at 24 weeks post-intervention between the groups, an analysis of covariance (ANCOVA) model will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm